CLINICAL TRIAL: NCT01326039
Title: Does Ultrasound-guided Ilioinguinal-iliohypogastric Block Improve Postoperative Pain Outcome After Unilateral Inguinal Hernia Repair?
Brief Title: Ultrasound-guided Ilioinguinal-iliohypogastric Block for Inguinal Hernia Repair
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Finn Bærentzen, MD, Copenhagen University Hospital Bispebjerg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBH_2010_IIH
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2010-04

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bupivacaine (Active Comparator): perineural bupivacaine 5 mg/ml 20 ml
  Interventions: Drug: bupivacaine
- saline (Placebo Comparator): perineural isotonic saline 20 ml
  Interventions: Drug: saline

INTERVENTIONS:
Drug: bupivacaine — perineural bupivacaine 5 mg/ml 20 ml
  Arms: bupivacaine
Drug: saline — perineural isotonic saline 20 ml
  Arms: saline

SUMMARY:
Aim: To investigate whether ultrasound-guided perineural administration of 20 ml bupivacaine 5 mg/ml vs 20 ml isotonic saline at the ilioinguinal-iliohypogastric nerves have a clinically analgesic effect after unilateral open inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* unilateral primary inguinal repair
* open surgery a.m. Lichtenstein
* informed consent

Exclusion Criteria:

* age below 18 years
* secondary surgery
* laparoscopic surgery
* lack of communicative skills

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
pain at mobilization using 100 mm VAS | within the first 24 hours postoperatively

SECONDARY OUTCOMES:
pain at rest using 100 mm VAS | within 24 hours postoperatively
perceived illness | within 24 hours postoperatively
  using short form-8 index
ability of daily living | within 24 hours
  using the Barthel/100 index
amount of analgesics | within 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jensen, MD, Study Chair — Copenhagen University Hospital Bispebjerg, Denmark
Locations (1):
- Copenhagen University Hospital Bispebjerg, Copenhagen, NV, Denmark